CLINICAL TRIAL: NCT06655870
Title: A Phase 1, Single-Center, Open-label, Single Ascending Dose and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Effects of mRNA-0184 Administered Subcutaneously in Healthy Participants
Brief Title: A Study to Investigate Safety and Tolerability of mRNA-0184 Administered Subcutaneously in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: mRNA-CRTX-002
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: mRNA-0184; Messenger RNA; Moderna

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD): mRNA-0184 (Experimental): Participants will receive a single subcutaneous (SC) injection of a fixed dose of mRNA-0184 on Day 1.
  Interventions: Drug: mRNA-0184
- Multiple Ascending Dose (MAD): mRNA-0184 (Experimental): Participants will receive up to 2 SC injections of a fixed dose of mRNA-0184 on Days 1 and 15.
  Interventions: Drug: mRNA-0184

INTERVENTIONS:
Drug: mRNA-0184 — SC injection

SUMMARY:
The purpose of this study is to test the safety of mRNA-0184 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, electrocardiogram (ECG), and vital signs.
* Body weight within 50 to 100 kilograms (kg) (inclusive) and body mass index within 18 to 32 kg/square meter (m^2) (inclusive) at Screening.
* Participant who could become pregnant must meet conditions as defined in the protocol.

Exclusion Criteria:

* History of any clinically significant disease or disorder, including bleeding disorders and wound healing disorders, which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
* Any clinically significant illness, or medical/surgical procedure, within 4 weeks of the first administration of the study drug (mRNA-0184).
* Any clinically significant abnormalities in clinical laboratory results at Screening. Repeat assessments are allowed at the Investigator's discretion if a false positive is suspected.
* Clinically significant abnormal findings in vital signs at Screening.
* Any positive result at Screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody.
* Use of any prescribed medication or over-the-counter (OTC) medication that may have an impact on the interpretation of study analyses in the opinion of the Investigator during the 2 weeks or 5 half-lives of the medication, whichever is longer, prior to the first administration of the study drug. Such prescribed or OTC medications are also not permitted during participation in the study. Hormonal contraception is permitted.
* Participation in another clinical study of another drug product (DP) within 30 days before Screening or within 5 terminal half-lives of the DP, whichever is longer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) Including Injection Site Reactions (ISRs), Adverse Events of Special Interests (AESIs), and Serious Adverse Events (SAEs) | Day 1 through Day 50

SECONDARY OUTCOMES:
Serum Concentrations of Study Drug | Day 1 through Day 50
Maximum Observed Plasma Concentration (Cmax) of Study Drug | Day 1 through Day 50
Area Under the Concentration-time Curve from Time 0 to Last Quantifiable Concentration (AUC0-t) of Study Drug | Day 1 through Day 50
Serum Concentrations of Relaxin-2-variable Light Chain Kappa (Rel2- vlk) Protein | Day 1 through Day 50
Maximum Observed Response (Emax) of Rel2- vlk Protein | Day 1 through Day 50
Area Under the Effect-time Curve (AUEC) of of Rel2- vlk Protein | Day 1 through Day 50
Number of Participants with Anti-Polyethylene Glycol (PEG) Antibodies | Day 1 through Day 50
Number of Participants with Anti-Rel2-vlk Protein Antibodies | Day 1 through Day 50

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia